CLINICAL TRIAL: NCT02975336
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study To Evaluate the Safety and Efficacy of M2951 in Subjects With SLE
Brief Title: A Phase II Study of M2951 in SLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is completed; primary analysis completed.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200527-0018; 2016-002950-19 (EudraCT Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; M2951; Placebo; Dose response; Oral Corticosteroids; Safety; Efficacy; Autoimmune And Inflammatory Disorders
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — evobrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Double-Blind Placebo-Controlled (DBPC) Period: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DBPC Period: M2951 25 mg QD (Experimental)
  Interventions: Drug: M2951
- DBPC Period: M2951 75 mg QD (Experimental)
  Interventions: Drug: M2951
- DBPC Period: M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951
- Long-Term Extension (LTE) Period: Placebo/ M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951
- LTE Period: M2951 25 mg QD/ M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951
- LTE Period: M2951 75 mg QD/ M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951
- LTE Period: M2951 50 mg BID/ M2951 50 mg BID (Experimental)
  Interventions: Drug: M2951

INTERVENTIONS:
Drug: Placebo — Participants received placebo matched to M2951 orally for 52 weeks.
  Arms: Double-Blind Placebo-Controlled (DBPC) Period: Placebo
Drug: M2951 — Participants received 25 milligrams (mg) of M2951 orally once daily (QD) for 52 weeks.
  Other Names: Evobrutinib
  Arms: DBPC Period: M2951 25 mg QD
Drug: M2951 — Participants received 75 mg of M2951 orally QD for 52 weeks.
  Other Names: Evobrutinib
  Arms: DBPC Period: M2951 75 mg QD
Drug: M2951 — Participants received 50 mg of M2951 orally twice daily (BID) for 52 weeks.
  Other Names: Evobrutinib
  Arms: DBPC Period: M2951 50 mg BID
Drug: M2951 — Participants who had received Placebo or M2951 (25 mg QD, 75 mg QD or 50 mg BID) during DBPC period were switched to receive 50 mg M2951 orally BID in LTE period for 104 weeks.
  Other Names: Evobrutinib
  Arms: LTE Period: M2951 25 mg QD/ M2951 50 mg BID; LTE Period: M2951 50 mg BID/ M2951 50 mg BID; LTE Period: M2951 75 mg QD/ M2951 50 mg BID; Long-Term Extension (LTE) Period: Placebo/ M2951 50 mg BID

SUMMARY:
M2951 is an investigational drug under evaluation for treatment of autoimmune and inflammatory disorders. The purpose of the study was to assess the Safety and Efficacy of M2951 in participants with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Eligible male and female participants, aged 18 to 75 years
* Must have diagnosis of SLE with either the Systemic Lupus International Collaborating Clinics (SLICC) criteria for SLE, or at least four of the 11 American College of Rheumatology (ACR) classification criteria for SLE, of at least six months duration prior to Screening
* SLEDAI-2K total score greater than or equal to (>=) 6 (including clinical SLEDAI greater than or equal to (>=) 4) at Screening Visit
* And be positive for anti-double-stranded Deoxyribonucleic Acid (DNA) and/or anti-nuclear antibody (ANA greater than or equal to (>=) 1:80) and/or anti-Smith (anti-Sm) antibody at the time of Screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants are not eligible for this study if they have active, clinically significant interstitial lung disease or pulmonary arterial hypertension
* Proteinuria (urine protein to creatinine ratio [UPCR] > 4 mg/mg)
* Acutely worsened renal function
* Central nervous system SLE
* Or within two weeks prior to Screening or during Screening: use of oral corticosteroids greater than (>) 30 mg daily prednisone equivalent
* Use of injectable corticosteroids, or change in dose of corticosteroids.
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (157):
- United States (42):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Medvin Clinical Research, Covina, California
  - Southern California Permanent Medical Group, Fontana, California
  - Global Research Management, Glendale, California
  - University of Southern California, Los Angeles, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Nazanin Firooz, MD Inc., West Hills, California
  - University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado
  - Yale School Of Medicine, New Haven, Connecticut
  - Clinical Research of West Florida - Corporate, Clearwater, Florida
  - Omega Research Consultants, DeBary, Florida
  - Center for Rheumatology, Immunology & Arthritis, Fort Lauderdale, Florida
  - Hope Clinical Trials, Miami, Florida
  - IRIS Research and Development, Plantation, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - Meridien Research, Inc., Tampa, Florida
  - Marietta Rheumatology Associates, PC, Marietta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - LSU Health Sciences Center Gastroenterology, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - AA MRC LLC Ahmed Arif Medical Research Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Innovative Clinical Research, LLC, Greenville, South Carolina
  - Metroplex Clinical Research Center, LLC, Dallas, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Accurate Clinical Management - Brionez, Houston, Texas
  - Medical Center Research, LLC Webster Office, Pearland, Texas
  - DM Clinical Research, Tomball, Texas
  - FSAEI HE " First Moscow State Medical University n.a. I.M. Sechenov" of the MoH of the RF, Seattle, Washington
- Argentina (14):
  - Instituto de Investigaciones Clinicas, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Centro Integral de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Instituto de Reumatologia, Mendoza
  - Cordis S.A., Salta
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
- Bulgaria (7):
  - UMHAT "Pulmed" OOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - Medizinski Zentar-1-Sevlievo EOOD, Sevlievo
  - Medical Center "Excelsior", OOD, Sofia
  - Medical Center Comac Medical EOOD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
- Chile (6):
  - Corporacion de Beneficencia Osorno, Osorno
  - Centro de Estudios Reumatologicos, Santiago
  - Centro Medico Prosalud, Santiago
  - Interin, Santiago
  - Psicomedica Clinical and Research Group, Santiago
  - Quantum Research Santiago, Santiago
- Colombia (5):
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla
  - Clínica de la Costa Ltda., Barranquilla
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogotá
  - Simedics Ips Sas, Bogotá
  - Servimed S.A.S., Bucaramanga
- Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin, Germany
- Italy (5):
  - Humanitas Research Hospital, Rozzano, Milano
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (15):
  - Ehime University Hospital, Toon-shi, Ehime
  - Tobata General Hospital, Kitakyushu-shi, Fukuoka
  - University of Occupational and Environmental Health Hospital, Kitakyushu-shi, Fukuoka
  - NHO Asahikawa Medical Center, Asahikawa-shi, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Eiraku Clinic, Kagoshima, Kagoshima-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - St. Luke's International Hospital, Chūōku, Tokyo-To
  - Tokyo Metropolitan Tama Medical Center, Fuchu-shi, Tokyo-To
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
  - Tottori University Hospital, Yonago-shi, Tottori
- Malaysia (5):
  - Hospital Pakar Sultanah Fatimah, Muar town, Johor
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
  - International Medical University (IMU) Healthcare, Bukit Jalil, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
- CAP Research, Solferino-Phoenix, Mauritius
- Mexico (9):
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas SC, Guadalajara, Jalisco
  - Unidad de Investigacion de las Enfermedades Reumaticas, Cuauhtémoc, Mexico City
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City, San Luis Potos
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
- Peru (9):
  - Hogar Clínica San Juan de Dios - Arequipa, Arequipa
  - Clinica El Golf, Lima
  - Clinica Medica Cayetano Heredia, Lima
  - Clinica San Juan Bautista, Lima
  - Clinica Vesalio, Lima
  - GINOBS SA. Instituto de Ginecologia y Reproduccion, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - University of Washington Medical Center, Lima
  - ICCV Research Instituto del Cerebro y la Columna Vertebral, Miraflores
- Philippines (7):
  - Angeles University Foundation Medical Center, Angeles City, Pampanga
  - Mary Mediatrix Medical Center, Batangas
  - De La Salle University Medical Center, Dasmariñas City, Cavite
  - Davao Doctors Hospital, Davao City
  - Southern Philippines Medical Center, Davao City
  - Iloilo Doctors Hospital, Iloilo City
  - St. Luke's Medical Center, Quezon City
- Poland (6):
  - CERMED, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska lek. Barbara Bazela, Elblag
  - Centrum Medyczne Plejady, Krakow
  - Nzoz Atopia, Krakow
  - Rheuma Medicus Zaklad, Warsaw
- Romania (3):
  - Spitalul Clinic "Dr.I. Cantacuzino", Bucharest
  - Spitalul Clinic "Sf. Maria", Bucharest
  - S.C Mediab S.R.L, Târgu Mureş
- Russia (9):
  - LLC "Alliance Biomedical - Ural Group", Izhevsk
  - TSBIH "Krasnoyarsk Interdistrict Clinical Hospital of Emergency Medical Care n.a. N.S. Karpovich, Krasnoyarsk
  - HMA - Hospital Maria Auxiliadora, Moscow
  - Ultramed, Omsk
  - LLC Medical Sanitary Unit#157, Saint Petersburg
  - Research Institute of Emergency Medical Care, Saint Petersburg
  - SPb SBIH "Clinical Rheumatological Hospital # 25", Saint Petersburg
  - SIH "Saratov City Clinical Hospital # 12", Saratov
  - Nebbiolo LLC, Tomsk
- South Africa (3):
  - Wits Clinical Research, Johannesburg, Gauteng
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
  - Naidoo, A - Netcare Umhlanga Hospital, Durban
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Konkuk University Medical Center, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung

REFERENCES:
- [Derived] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Bolay CL, Kao AH, Guehring H. A plain language summary of what clinical studies can tell us about the safety of evobrutinib - a potential treatment for multiple sclerosis. Neurodegener Dis Manag. 2023 Aug;13(4):207-213. doi: 10.2217/nmt-2023-0003. Epub 2023 Jun 22. PMID 37345645
- [Derived] Montalban X, Wallace D, Genovese MC, Tomic D, Parsons-Rich D, Le Bolay C, Kao AH, Guehring H. Characterisation of the safety profile of evobrutinib in over 1000 patients from phase II clinical trials in multiple sclerosis, rheumatoid arthritis and systemic lupus erythematosus: an integrated safety analysis. J Neurol Neurosurg Psychiatry. 2023 Jan;94(1):1-9. doi: 10.1136/jnnp-2022-328799. Epub 2022 Nov 23. PMID 36418156
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527-0018
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1053 participants with Systemic Lupus Erythematosus (SLE) were screened. Out of which 469 participants were randomized in ratio of 1:1:1:1 to 1 of 4 treatment groups: Placebo; M2951 25mg QD, M2951 75 mg QD and M2951 50 mg BID. 283 out of 348 participants that completed Double-Blind Placebo-Controlled (DBPC) period, entered the Long-Term Extension (LTE) period of study.
Groups:
- DBPC Period: Placebo: Participants received placebo matched to M2951 orally for 52 weeks.
- DBPC Period: M2951 25 mg QD: Participants received 25 milligrams (mg) of M2951 orally once daily (QD) for 52 weeks.
- DBPC Period: M2951 75 mg QD: Participants received 75 mg of M2951 orally QD for 52 weeks.
- DBPC Period: M2951 50 mg BID: Participants received 50 mg of M2951 orally twice daily (BID) for 52 weeks.
- LTE: Placebo/ M2951 50 mg BID: Participants who received Placebo in DBPC period were switched to receive 50 mg M2951 orally BID in LTE period for 104 weeks.
- LTE Period: M2951 25 mg QD/ M2951 50 mg BID: Participants who received 25 mg of M2951 orally QD in DBPC period were switched to receive 50 mg M2951 orally BID in LTE period for 104 weeks.
- LTE Period: M2951 75 mg QD/ M2951 50 mg BID: Participants who received 75 mg of M2951 orally QD in DBPC period were switched to receive 50 mg M2951 orally BID in LTE period for 104 weeks.
- LTE: M2951 50 mg BID/ M2951 50 mg BID: Participants who received 50 mg of M2951 orally BID in DBPC period continued to receive same dose of M2951 orally BID in LTE period for 104 weeks.
Period: DBPC (52 Weeks)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID | LTE: Placebo/ M2951 50 mg BID | LTE Period: M2951 25 mg QD/ M2951 50 mg BID | LTE Period: M2951 75 mg QD/ M2951 50 mg BID | LTE: M2951 50 mg BID/ M2951 50 mg BID
Started | 117 | 118 | 117 | 117 | 0 | 0 | 0 | 0
Completed | 85 | 89 | 90 | 84 | 0 | 0 | 0 | 0
Not Completed | 32 | 29 | 27 | 33 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 16 | 17 | 13 | 18 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 4 | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Premature termination of the study | 5 | 6 | 6 | 4 | 0 | 0 | 0 | 0
Period: LTE (104 Weeks)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID | LTE: Placebo/ M2951 50 mg BID | LTE Period: M2951 25 mg QD/ M2951 50 mg BID | LTE Period: M2951 75 mg QD/ M2951 50 mg BID | LTE: M2951 50 mg BID/ M2951 50 mg BID
Started | 0 | 0 | 0 | 0 | 62 | 69 | 80 | 72
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 62 | 69 | 80 | 72
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 7 | 4 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 55 | 63 | 76 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID | Total
Number analyzed (Participants) | 117 | 118 | 117 | 117 | 469
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (12.49) | 38.8 (12.45) | 41.5 (12.52) | 42.2 (11.78) | 40.7 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 112 | 111 | 112 | 445
  Male | 7 | 6 | 6 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 51 | 47 | 42 | 185
  Not Hispanic or Latino | 72 | 67 | 70 | 75 | 284
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 23 | 17 | 21 | 13 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 11 | 12 | 45
  White | 66 | 73 | 68 | 83 | 290
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 18 | 16 | 17 | 9 | 60

OUTCOME MEASURES:

1. Primary Outcome: DBPC Period: Number of Participants With Response Based on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Week 52
Description: SRI-4 response was defined as greater than or equal to (>=) 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score, no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and no treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to Systemic Lupus Erythematosus (SLE) divided into 9 organ systems. For each organ system A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale =from 0(very well) to 100(very poor).
Time Frame: Week 52
Population: The modified Intent To Treat (mITT) analysis set included all randomized participants who had received at least one dose of Investigational Medicinal Product (IMP) [Evobrutinib or placebo] and have at least one Baseline and one post Baseline disease assessment (among the following: Systemic Lupus Erythematosus Disease Activity Index flare index [SFI], SLEDAI 2K, PGA, BILAG 2004, Cutaneous Lupus Erythematosus Disease Area and Severity Index [CLASI]).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants | 52 | 64 | 60 | 55
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.91 to 2.64]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.76 to 2.18]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.67 to 1.93]

2. Primary Outcome: DBPC Period: Number of Participants With Response Based on Systemic Lupus Erythematosus Responder Index 6 (SRI-6) at Week 52
Description: SRI-6 response was defined as >= 6-point reduction in SLEDAI-2K total score, no new BILAG A and no more than 1 new BILAG B domain score and no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system :A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale =from 0(very well) to 100(very poor).
Time Frame: Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "overall number of participants analyzed" signifies those participants who achieved SLEDAI-2K total score >= 10 at screening (High Disease Activity [HDA] participants).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 56 | 54 | 65 | 55
Participants | 22 | 27 | 30 | 24
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.69 to 3.24]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.68 to 2.97]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.59 to 2.75]

3. Primary Outcome: DBPC Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs: events between first dose of study drug that were absent before treatment/that worsened relative to pre-treatment state up to 56 weeks. TEAEs included both serious TEAEs and non-serious TEAEs. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: Baseline up to Week 56
Population: The safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 117 | 118 | 117 | 117
Participants
  Any TEAEs | 96 | 103 | 100 | 99
  Any serious TEAE | 10 | 13 | 11 | 9

4. Primary Outcome: DBPC Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Severity of TEAEs were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 1= Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with TEAEs by severity were reported.
Time Frame: Baseline up to Week 56
Population: The Safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 117 | 118 | 117 | 117
Participants
  Grade 1 | 76 | 80 | 79 | 76
  Grade 2 | 63 | 77 | 72 | 78
  Grade 3 | 24 | 29 | 24 | 21
  Grade 4 | 1 | 1 | 0 | 2
  Grade 5 | 0 | 1 | 1 | 0

5. Primary Outcome: DBPC Period: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure, pulse rate, respiratory rate, weight and height. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in vital signs were reported.
Time Frame: Baseline up to Week 56
Population: The safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 117 | 118 | 117 | 117
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: DBPC Period: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. The corrected QT interval (QTcF) was calculated using Fridericia's formula. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: Baseline up to Week 56
Population: The safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 117 | 118 | 117 | 117
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: DBPC Period: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry, urinalysis and coagulation. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Time Frame: Baseline up to Week 56
Population: The safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 117 | 118 | 117 | 117
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 2
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 2.
Time Frame: Week 2
Population: The Safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 116 | 115 | 113
gram per liter (g/L)
  IgG | 14.56 (5.367) | 13.75 (4.652) | 14.37 (5.536) | 12.81 (3.847)
  IgA | 2.62 (1.207) | 2.75 (1.374) | 2.78 (1.328) | 2.66 (1.137)
  IgM | 1.12 (0.662) | 1.22 (0.890) | 1.09 (0.697) | 1.18 (0.776)

9. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 4
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 4.
Time Frame: Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 114 | 114 | 115
gram per liter (g/L)
  IgG | 14.92 (5.497) | 13.60 (4.590) | 14.21 (4.828) | 12.73 (3.771)
  IgA | 2.71 (1.284) | 2.73 (1.349) | 2.82 (1.293) | 2.64 (1.109)
  IgM | 1.12 (0.699) | 1.18 (0.824) | 1.06 (0.676) | 1.16 (0.745)

10. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 12
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 12.
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 106 | 110 | 105
gram per liter (g/L)
  IgG: | 14.91 (5.312) | 12.92 (4.332) | 13.64 (4.035) | 12.38 (3.520)
  IgA | 2.72 (1.321) | 2.73 (1.340) | 2.88 (1.363) | 2.68 (1.021)
  IgM | 1.11 (0.683) | 1.05 (0.700) | 0.95 (0.610) | 1.02 (0.695)

11. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 24
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 24.
Time Frame: Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 101 | 96
gram per liter (g/L)
  IgG | 15.01 (5.190) | 13.75 (4.783) | 13.79 (4.165) | 12.86 (3.725)
  IgA | 2.79 (1.430) | 2.89 (1.460) | 2.98 (1.391) | 2.78 (1.091)
  IgM | 1.07 (0.609) | 1.01 (0.686) | 0.89 (0.583) | 0.98 (0.656)

12. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 36
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 36.
Time Frame: Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 92 | 91 | 97 | 86
gram per liter (g/L)
  IgG | 14.81 (5.217) | 13.54 (4.242) | 13.67 (3.934) | 12.65 (3.480)
  IgA | 2.72 (1.378) | 2.89 (1.418) | 3.01 (1.420) | 2.86 (1.073)
  IgM | 1.06 (0.630) | 1.01 (0.669) | 0.85 (0.541) | 0.95 (0.656)

13. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 52
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 52
Time Frame: Week 52
Population: The Safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 78 | 83 | 85 | 76
gram per liter (g/L)
  IgG | 15.21 (5.105) | 13.90 (4.087) | 14.32 (4.542) | 13.01 (3.723)
  IgA | 2.82 (1.438) | 2.95 (1.596) | 3.17 (1.596) | 2.95 (1.159)
  IgM: number analyzed (Participants) | 78 | 83 | 84 | 76
  IgM | 1.08 (0.624) | 0.94 (0.645) | 0.82 (0.487) | 0.96 (0.670)

14. Primary Outcome: DBPC Period: Mean Absolute Value of Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 56
Description: Mean absolute value of serum levels of IgG, IgA, IgM were assessed at Week 56
Time Frame: Week 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 37 | 36 | 31 | 33
gram per liter (g/L)
  IgG | 14.82 (5.504) | 14.25 (4.435) | 14.25 (4.626) | 13.12 (4.507)
  IgA | 2.95 (1.549) | 3.01 (1.459) | 2.89 (1.655) | 3.03 (1.164)
  IgM | 1.11 (0.642) | 1.01 (0.601) | 0.95 (0.624) | 1.31 (0.869)

15. Primary Outcome: DBPC Period: Mean Absolute Total B Cell Count at Week 4
Description: Mean total B cell count were assessed. Flow cytometry analysis of lymphocyte populations using four-color fluorescence activated cell sorting was performed for the analysis of B cell counts.
Time Frame: Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 98 | 99 | 99 | 99
Cells per microliter | 150 (126.9) | 236 (197.4) | 296 (243.8) | 229 (232.9)

16. Primary Outcome: DBPC Period: Mean Absolute Total B Cell Count at Week 24
Description: Mean absolute total B cell count were assessed. Flow cytometry analysis of lymphocyte populations using four-color fluorescence activated cell sorting was performed for the analysis of B cell counts.
Time Frame: Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 89 | 90 | 87 | 88
Cells per microliter | 161 (125.8) | 184 (152.6) | 204 (158.3) | 151 (129.2)

17. Primary Outcome: DBPC Period: Mean Absolute Total B Cell Count at Week 52
Description: as for outcome 16
Time Frame: Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 68 | 66 | 76 | 66
Cells per microliter | 169 (121.9) | 167 (168.7) | 180 (170.7) | 119 (84.1)

18. Primary Outcome: DBPC Period: Mean Absolute Total B Cell Count at Week 56
Description: as for outcome 16
Time Frame: Week 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 35 | 30 | 27 | 30
Cells per microliter | 164 (113.3) | 129 (100.0) | 156 (127.1) | 104 (71.9)

19. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 2
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 116 | 115 | 113
gram per liter (g/L)
  IgG | -0.51 (1.726) | -0.06 (1.361) | -0.15 (1.772) | -0.40 (1.025)
  IgA | -0.11 (0.435) | -0.04 (0.431) | -0.01 (0.381) | -0.03 (0.268)
  IgM | 0.00 (0.197) | -0.05 (0.194) | -0.04 (0.155) | -0.07 (0.116)

20. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 4
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 114 | 114 | 115
gram per liter (g/L)
  IgG | -0.26 (1.760) | -0.16 (1.463) | -0.24 (1.657) | -0.45 (1.150)
  IgA | -0.01 (0.205) | -0.04 (0.334) | 0.03 (0.447) | -0.03 (0.301)
  IgM | 0.01 (0.195) | -0.09 (0.175) | -0.07 (0.192) | -0.08 (0.159)

21. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 12
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 106 | 110 | 105
gram per liter (g/L)
  IgG | -0.36 (2.073) | -0.62 (1.827) | -0.72 (2.552) | -0.93 (1.640)
  IgA | 0.00 (0.325) | -0.02 (0.360) | 0.06 (0.518) | -0.03 (0.340)
  IgM | -0.01 (0.194) | -0.20 (0.301) | -0.18 (0.277) | -0.20 (0.250)

22. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 24
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 96 | 97 | 101 | 96
gram per liter (g/L)
  IgG | -0.21 (2.318) | 0.11 (2.234) | -0.46 (2.912) | -0.57 (2.363)
  IgA | 0.06 (0.332) | 0.14 (0.390) | 0.19 (0.565) | 0.04 (0.563)
  IgM | -0.01 (0.264) | -0.23 (0.369) | -0.23 (0.321) | -0.25 (0.346)

23. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 36
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 92 | 91 | 97 | 86
gram per liter (g/L)
  IgG | -0.15 (2.130) | 0.02 (2.487) | -0.43 (2.572) | -0.69 (2.189)
  IgA | -0.02 (0.361) | 0.22 (0.453) | 0.24 (0.583) | 0.08 (0.459)
  IgM | -0.04 (0.255) | -0.25 (0.416) | -0.25 (0.284) | -0.28 (0.392)

24. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 52
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 52
Population: The Safety analysis set included all participants who received at least 1 dose of IMP (Evobrutinib or Placebo). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 78 | 83 | 85 | 76
gram per liter (g/L)
  IgG | 0.41 (2.898) | 0.29 (2.361) | 0.35 (2.688) | -0.31 (2.344)
  IgA | 0.19 (0.420) | 0.32 (0.492) | 0.39 (0.767) | 0.18 (0.469)
  IgM: number analyzed (Participants) | 78 | 83 | 84 | 76
  IgM | -0.02 (0.235) | -0.25 (0.303) | -0.21 (0.318) | -0.33 (0.456)

25. Primary Outcome: DBPC Period: Change From Baseline in Serum Immunoglobulin (Ig) Levels (IgG, IgA, IgM) at Week 56
Description: Change from baseline in the serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline and Week 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 37 | 36 | 31 | 33
gram per liter (g/L)
  IgG | 0.74 (2.907) | 1.06 (2.607) | 0.74 (1.987) | -0.40 (2.823)
  IgA | 0.23 (0.468) | 0.48 (0.600) | 0.35 (0.488) | 0.26 (0.498)
  IgM | 0.01 (0.266) | -0.15 (0.219) | -0.11 (0.225) | -0.21 (0.488)

26. Primary Outcome: DBPC Period: Change From Baseline in Total B Cell Count at Week 4
Description: Change from baseline in Total B cell count were assessed. Flow cytometry analysis of lymphocyte populations using four-color fluorescence-activated cell sorting was performed for the analysis of B cell counts.
Time Frame: Baseline and Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 90 | 88 | 88 | 91
Cells per microliter | -5 (93.7) | 65 (146.6) | 87 (146.2) | 67 (109.1)

27. Primary Outcome: DBPC Period: Change From Baseline in Total B Cell Count at Week 24
Description: as for outcome 26
Time Frame: Baseline and Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 80 | 82 | 73 | 81
Cells per microliter | 2 (98.1) | 5 (112.0) | 3 (103.2) | -7 (134.7)

28. Primary Outcome: DBPC Period: Change From Baseline in Total B Cell Count at Week 52
Description: as for outcome 26
Time Frame: Baseline and Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 57 | 60 | 63 | 60
Cells per microliter | -14 (103.0) | -19 (133.3) | -14 (147.5) | -52 (215.7)

29. Primary Outcome: DBPC Period: Change From Baseline in Total B Cell Count at Week 56
Description: as for outcome 26
Time Frame: Baseline and Week 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 30 | 27 | 24 | 24
Cells per microliter | 7 (96.2) | -70 (138.2) | -75 (192.1) | -48 (85.8)

30. Secondary Outcome: DBPC Period: Time to First Severe British Isles Lupus Assessment Group (BILAG) A Flare
Description: BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system based on alphabetic score: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. BILAG evaluated by scoring each of a list of signs and symptoms as: improving (1); same (2); worse (3); new (4); not present (0); not done (ND). Total BILAG score is sum of scores of 9 domains where A=12, B=8, C=1, D=0, and E=0. Total score ranges from 0 to 108 with a higher score indicating greater lupus activity. Time to first severe flare, where a severe flare is defined as at least one BILAG A (Severe disease activity) score in any organ system due to items that are new or worse, compared to the BILAG evaluation at the previous visit, during the 52-Week Treatment. It was measured using Kaplan-Meier (KM) estimates.
Time Frame: Baseline up to Week 56
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 14 | 16 | 11 | 12
Days | NA [29.0 to 337.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [29.0 to 367.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [29.0 to 225.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [28.0 to 162.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value.
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.7034, Cox proportional hazards model; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.57 to 2.40]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.5462, Cox proportional hazards model; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.31 to 1.52]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5462, Cox proportional hazards model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.42 to 1.97]

31. Secondary Outcome: DBPC Period: Number of Participants With Response Based on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Week 52 in Serologically Active (SA) Subgroup
Description: SRI-4 response was defined as greater than or equal to (>=) 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score, no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and no treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to Systemic Lupus Erythematosus (SLE), divided into 9 organ systems. For each organ system A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale =from 0(very well) to 100(very poor).
Time Frame: Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "Overall Number of Participants Analyzed" signifies those participants with positive anti-double-stranded deoxyribonucleic acid (antidsDNA) and/or low complement levels at screening (Serologically active subgroup).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 59 | 65 | 60 | 63
Participants | 28 | 38 | 29 | 34
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.74 to 3.15]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.49 to 2.13]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5462, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.65 to 2.81]

32. Secondary Outcome: DBPC Period: Number of Participants With Response Based on Systemic Lupus Erythematosus Responder Index 6 (SRI-6) at Week 52 in Serologically Active Subgroup
Description: SRI-6 response was defined as >= 6-point reduction in SLEDAI-2K total score, no new BILAG A and no more than 1 new BILAG B domain score and no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system :A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale = from 0(very well) to 100(very poor).
Time Frame: Week 52
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 59 | 65 | 60 | 63
Participants | 17 | 25 | 23 | 23
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.2434, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.73 to 3.54]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.2389, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.73 to 3.63]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.1952, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.76 to 3.85]

33. Secondary Outcome: DBPC Period: Time to First British Isles Lupus Assessment Group (BILAG) A or 2B Moderate to Severe Flare
Description: BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system based on alphabetic score: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. BILAG evaluated by scoring each of a list of signs and symptoms as: improving (1); same (2); worse (3); new (4); not present (0); not done (ND). Total BILAG score is sum of scores of 9 domains where A=12, B=8, C=1, D=0, and E=0. Total score ranges from 0 to 108 with a higher score indicating greater lupus activity. A Moderate to Severe (BILAG A or 2B) flare is defined as at least one BILAG A (severe disease activity) grade or two BILAG B (moderate disease activity) grade in any organ system due to items that are new or worse, compared to the BILAG evaluation at the previous visit, during the 52 week treatment. It was measured using Kaplan-Meier (KM) estimates.
Time Frame: Baseline up to Week 56
Population: as for outcome 30
Measure: Median (Full Range); unit: Days
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 18 | 27 | 19 | 19
Days | NA [29.0 to 337.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [27.0 to 365.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [29.0 to 308.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value. | NA [28.0 to 334.0] — NA indicated that median was not reached as the number of participants with events were too low in respect to number of participants censored to estimate the value.
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.0987, Cox proportional hazards model; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.87 to 2.89]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.9201, Cox proportional hazards model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.51 to 1.85]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5645, Cox proportional hazards model; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.60 to 2.20]

34. Secondary Outcome: DBPC Period: Number of Participants With British Isles Lupus Assessment Group (BILAG) 2004 Flare-Free Status During the 52-Week Treatment Period
Description: A participant has a flare-free status if no flare has been reported during the 52-week treatment period. Participants who discontinued treatment prior to Week 52, without having a flare are counted as not being flare free at Week 52. A flare was defined as either 1 or more new BILAG-2004 A (severe disease activity) or 2 or more new BILAG-2004 B (moderate disease activity) items compared to the previous visit. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system based on alphabetic score: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected.
Time Frame: up to Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI.
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants | 41 | 35 | 37 | 33
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.3743, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.44 to 1.37]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.6445, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.50 to 1.54]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.2634, Regression, Logistic; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.41 to 1.28]

35. Secondary Outcome: DBPC Period: Annualized Flare Rate
Description: A flare was defined as either 1 or more new BILAG-2004 A (severe disease activity) or 2 or more new BILAG-2004 B (moderate disease activity) items compared to the previous visit. The occurrence of a new flare was checked for each available visit versus the previous available visit up to Week 52. If no new flares occurred, the number of flares was set to 0. Otherwise all flares were counted leading to the maximum number of flares of 13. The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days multiplied with 365.25 (1 year). The flare exposure time is the time up to Week 52 (date of BILAG-2004 assessment at Week 52) or up to the date of last available BILAG 2004 assessment.
Time Frame: Baseline up to Week 52
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Annualized flare rate ratio
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Annualized flare rate ratio | 0.15 [0.06 to 0.39] | 0.23 [0.09 to 0.59] | 0.13 [0.05 to 0.33] | 0.19 [0.07 to 0.51]
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.2989, Negative binomial regression — Nominal p-value; Rate Ratio = 1.59, 95% CI 2-sided [0.66 to 3.81]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.7325, Negative binomial regression — Nominal p-value; Rate Ratio = 0.85, 95% CI 2-sided [0.33 to 2.19]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5910, Negative binomial regression — Nominal p-value; Rate Ratio = 1.29, 95% CI 2-sided [0.51 to 3.22]

36. Secondary Outcome: DBPC Period: Number of Participants With Low Disease Activity Status, Defined by Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) Score of Less Than or Equal (<= ) 2 at Week 52
Description: Low disease activity is defined as SLEDAI-2K score <=2. SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 30 days. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: Week 52
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants | 26 [15.5 to 31.6] | 32 [19.9 to 37.0] | 39 [25.1 to 43.0] | 28 [17.0 to 33.5]
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.3635, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.72 to 2.47]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.0329, Regression, Logistic; Odds Ratio (OR) = 1.94, 95% CI 2-sided [1.06 to 3.56]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.7619, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.59 to 2.07]

37. Secondary Outcome: DBPC Period: Number of Participants With Low Disease Activity Status, Defined by Clinical Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) Score of Less Than or Equal (<= ) 2 at Week 52
Description: Low disease activity is defined as SLEDAI-2K score <=2. SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 30 days. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms). Clinical SLEDAI-2K score is equal to the SLEDAI-2K score from electronic case report form (eCRF) excluding the components 'Increased Deoxyribonucleic acid (DNA) Binding' and 'Low Complement'.
Time Frame: Week 52
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants | 42 [28.0 to 46.4] | 50 [34.3 to 53.0] | 52 [35.6 to 54.3] | 41 [27.2 to 45.5]
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.2642, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.79 to 2.35]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.1489, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.87 to 2.57]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.9285, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.56 to 1.70]

38. Secondary Outcome: DBPC Period: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) Score at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 30 days. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: The mITT analysis set included all randomized participants who had received at least 1 dose of IMP (Evobrutinib or placebo) and have at least 1 Baseline and 1 post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 111 | 115 | 115 | 113
Units on a Scale
  Week 4 | -1 (1.9) | -1 (2.1) | 0 (1.9) | -1 (2.2)
  Week 8: number analyzed (Participants) | 111 | 111 | 112 | 109
  Week 8 | -2 (3.1) | -2 (3.2) | -2 (3.0) | -2 (3.2)
  Week 12: number analyzed (Participants) | 109 | 106 | 109 | 104
  Week 12 | -3 (3.8) | -3 (3.3) | -3 (3.2) | -3 (3.4)
  Week 16: number analyzed (Participants) | 104 | 102 | 107 | 98
  Week 16 | -4 (3.7) | -3 (3.4) | -3 (3.4) | -3 (3.6)
  Week 20: number analyzed (Participants) | 101 | 99 | 103 | 96
  Week 20 | -4 (4.1) | -4 (3.8) | -4 (3.4) | -4 (3.4)
  Week 24: number analyzed (Participants) | 98 | 95 | 101 | 94
  Week 24 | -4 (4.0) | -4 (3.7) | -4 (3.6) | -3 (3.4)
  Week 28: number analyzed (Participants) | 93 | 94 | 99 | 89
  Week 28 | -4 (3.9) | -4 (3.6) | -4 (3.5) | -4 (3.5)
  Week 32: number analyzed (Participants) | 92 | 91 | 97 | 88
  Week 32 | -4 (4.0) | -4 (3.5) | -4 (3.7) | -4 (3.4)
  Week 36: number analyzed (Participants) | 91 | 90 | 95 | 113
  Week 36 | -4 (4.3) | -5 (3.5) | -5 (3.6) | -4 (3.5)
  Week 40: number analyzed (Participants) | 90 | 90 | 95 | 87
  Week 40 | -5 (4.1) | -5 (3.6) | -5 (3.8) | -4 (3.3)
  Week 44: number analyzed (Participants) | 89 | 90 | 92 | 86
  Week 44 | -4 (4.0) | -5 (3.7) | -5 (3.9) | -4 (3.5)
  Week 48: number analyzed (Participants) | 89 | 90 | 92 | 85
  Week 48 | -4 (4.1) | -5 (3.7) | -5 (3.8) | -5 (3.3)
  Week 52: number analyzed (Participants) | 85 | 89 | 91 | 84
  Week 52 | -5 (4.0) | -5 (3.7) | -5 (3.7) | -5 (3.9)

39. Secondary Outcome: DBPC Period: Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: CLASI is an validated measurement instrument for lupus erythematosus developed for use in clinical studies that consists of separate scores for the activity of the disease (CLASI-A). The CLASI activity score is calculated on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. The CLASI activity score ranges from 0-70, with higher scores indicating more severe skin disease. Severity categories based on the CLASI activity score are as follows: mild (0-9), moderate (10-20), and severe (21-70).
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 111 | 113 | 115 | 113
Units on a Scale
  Week 2: number analyzed (Participants) | 110 | 113 | 113 | 109
  Week 2 | -1 (1.9) | -1 (1.6) | 0 (1.6) | 0 (1.2)
  Week 4 | -1 (1.9) | -1 (3.5) | -1 (2.4) | -1 (2.2)
  Week 8: number analyzed (Participants) | 110 | 109 | 110 | 107
  Week 8 | -2 (2.8) | -1 (4.2) | -1 (2.3) | -1 (2.5)
  Week 12: number analyzed (Participants) | 107 | 104 | 107 | 101
  Week 12 | -2 (2.8) | -2 (3.3) | -2 (3.2) | -2 (2.7)
  Week 16: number analyzed (Participants) | 104 | 102 | 107 | 98
  Week 16 | -2 (3.1) | -2 (3.9) | -2 (3.3) | -2 (2.7)
  Week 20: number analyzed (Participants) | 99 | 96 | 102 | 95
  Week 20 | -3 (3.6) | -3 (4.4) | -3 (3.4) | -2 (2.9)
  Week 24: number analyzed (Participants) | 97 | 95 | 100 | 92
  Week 24 | -3 (3.5) | -3 (4.7) | -3 (3.6) | -2 (2.7)
  Week 28: number analyzed (Participants) | 92 | 91 | 96 | 89
  Week 28 | -3 (3.7) | -3 (4.6) | -3 (3.4) | -2 (2.7)
  Week 32: number analyzed (Participants) | 91 | 91 | 96 | 87
  Week 32 | -3 (3.5) | -3 (4.4) | -3 (3.6) | -3 (3.2)
  Week 36: number analyzed (Participants) | 90 | 89 | 95 | 86
  Week 36 | -3 (3.5) | -3 (4.6) | -3 (3.4) | -3 (3.6)
  Week 40: number analyzed (Participants) | 90 | 90 | 92 | 85
  Week 40 | -3 (3.0) | -3 (4.6) | -3 (3.6) | -3 (3.8)
  Week 44: number analyzed (Participants) | 89 | 90 | 92 | 85
  Week 44 | -3 (3.2) | -3 (4.5) | -3 (3.7) | -3 (3.8)
  Week 48: number analyzed (Participants) | 88 | 89 | 91 | 83
  Week 48 | -3 (3.2) | -3 (4.7) | -3 (3.7) | -3 (3.9)
  Week 52: number analyzed (Participants) | 84 | 86 | 89 | 84
  Week 52 | -3 (3.6) | -4 (4.8) | -3 (3.7) | -3 (4.0)

40. Secondary Outcome: DBPC Period: Number of Participants With Response Based on BILAG-Based Composite Lupus Assessment (BICLA) at Week 52
Description: BICLA response defined as participants meeting following criteria: [1] At least one gradation of improvement in baseline BILAG scores in all body systems with moderate or severe disease activity at entry (example: all A (severe disease) scores falling to B (moderate), C (mild), or D (no activity) and all B scores falling to C or D; [2] No new BILAG A or more than one new BILAG B scores; [3] No worsening of total SLEDAI-2K score from baseline; [4] No significant deterioration (=<10%) in physician's global assessment and [5] No treatment failure (initiation of non-protocol treatment).
Time Frame: Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "Overall Number of Participants Analyzed" signifies those participants who have at least 1 BILAG A or 2 BILAG B grades at Baseline (BICLA Subpopulation).
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 76 | 73 | 76 | 70
Participants | 30 | 29 | 33 | 24
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.9061, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.49 to 1.88]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.6053, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.61 to 2.31]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.5200, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.40 to 1.59]

41. Secondary Outcome: DBPC Period: Change From Baseline in British Isles Lupus Assessment Group (BILAG)-2004 Score at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: BILAG 2004 disease activity Index: assessing clinical signs, symptoms, or laboratory parameters related to SLE, divided into 9 organ systems. For each organ system based on alphabetic score: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. BILAG evaluated by scoring each of a list of signs and symptoms as: improving (1); same (2); worse (3); new (4); not present (0); not done (ND). Total BILAG score is sum of scores of 9 domains where A=12, B=8, C=1, D=0, and E=0. Total score ranges from 0 to 108 with a higher score indicating greater lupus activity.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 111 | 109 | 109
Units on a Scale
  Week 4: number analyzed (Participants) | 108 | 108 | 108 | 105
  Week 4 | -4 (5.8) | -4 (6.1) | -3 (6.3) | -4 (6.2)
  Week 8 | -6 (6.0) | -5 (7.0) | -6 (6.3) | -6 (6.1)
  Week 12: number analyzed (Participants) | 109 | 106 | 107 | 104
  Week 12 | -7 (6.7) | -7 (6.8) | -6 (7.0) | -6 (6.2)
  Week 16: number analyzed (Participants) | 104 | 102 | 105 | 98
  Week 16 | -7 (6.9) | -7 (7.6) | -6 (6.8) | -6 (5.9)
  Week 20: number analyzed (Participants) | 101 | 99 | 102 | 96
  Week 20 | -7 (6.8) | -7 (7.3) | -7 (7.6) | -6 (6.2)
  Week 24: number analyzed (Participants) | 97 | 95 | 100 | 94
  Week 24 | -8 (6.9) | -7 (6.5) | -8 (7.7) | -6 (6.3)
  Week 28: number analyzed (Participants) | 93 | 94 | 98 | 89
  Week 28 | -8 (6.7) | -8 (6.9) | -8 (7.4) | -7 (6.2)
  Week 32: number analyzed (Participants) | 92 | 91 | 96 | 89
  Week 32 | -9 (6.7) | -8 (7.3) | -8 (7.9) | -7 (6.0)
  Week 36: number analyzed (Participants) | 91 | 90 | 95 | 88
  Week 36 | -8 (7.1) | -8 (7.2) | -8 (7.4) | -7 (6.7)
  Week 40: number analyzed (Participants) | 88 | 90 | 95 | 87
  Week 40 | -9 (6.8) | -8 (6.7) | -9 (7.7) | -7 (6.6)
  Week 44: number analyzed (Participants) | 88 | 90 | 92 | 85
  Week 44 | -9 (7.2) | -9 (7.2) | -9 (7.9) | -7 (6.7)
  Week 48: number analyzed (Participants) | 89 | 90 | 92 | 85
  Week 48 | -8 (7.1) | -8 (7.2) | -9 (7.6) | -7 (6.5)
  Week 52: number analyzed (Participants) | 85 | 89 | 91 | 84
  Week 52 | -8 (7.0) | -9 (6.8) | -9 (7.8) | -7 (6.7)

42. Secondary Outcome: DBPC Period: Change From Baseline in Physician's Global Assessment (PGA) Score at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 millimeter horizontal Visual Analog Scale (VAS). Physician rated participant's disease activity on a scale ranged from 0-100 millimeter (mm), where 0 indicated no disease activity and 100 represented maximum disease activity.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 111 | 115 | 115 | 113
Millimeter
  Week 4 | -8 (11.7) | -8 (14.1) | -9 (13.4) | -9 (12.1)
  Week 8: number analyzed (Participants) | 110 | 109 | 111 | 107
  Week 8 | -13 (16.2) | -14 (16.5) | -13 (15.5) | -14 (15.9)
  Week 12: number analyzed (Participants) | 107 | 104 | 107 | 101
  Week 12 | -18 (17.4) | -18 (18.8) | -19 (18.3) | -18 (16.9)
  Week 16: number analyzed (Participants) | 104 | 102 | 105 | 98
  Week 16 | -21 (17.6) | -20 (19.7) | -21 (18.7) | -19 (18.0)
  Week 20: number analyzed (Participants) | 99 | 96 | 102 | 95
  Week 20 | -23 (19.2) | -21 (19.5) | -24 (17.9) | -20 (18.6)
  Week 24: number analyzed (Participants) | 97 | 95 | 100 | 92
  Week 24 | -24 (17.8) | -24 (20.0) | -25 (19.2) | -21 (18.0)
  Week 28: number analyzed (Participants) | 92 | 91 | 96 | 89
  Week 28 | -26 (17.6) | -26 (20.3) | -26 (18.6) | -24 (17.8)
  Week 32: number analyzed (Participants) | 91 | 91 | 96 | 87
  Week 32 | -26 (17.8) | -26 (20.8) | -26 (19.0) | -26 (17.5)
  Week 36: number analyzed (Participants) | 90 | 89 | 95 | 86
  Week 36 | -26 (17.9) | -26 (20.9) | -29 (18.3) | -26 (18.3)
  Week 40: number analyzed (Participants) | 90 | 90 | 91 | 85
  Week 40 | -27 (16.9) | -27 (19.1) | -30 (19.7) | -25 (18.1)
  Week 44: number analyzed (Participants) | 89 | 90 | 92 | 85
  Week 44 | -28 (16.6) | -28 (20.1) | -30 (20.7) | -26 (16.6)
  Week 48: number analyzed (Participants) | 88 | 89 | 91 | 83
  Week 48 | -29 (16.5) | -29 (19.5) | -32 (18.8) | -28 (18.3)
  Week 52: number analyzed (Participants) | 84 | 86 | 89 | 84
  Week 52 | -29 (16.2) | -31 (20.7) | -33 (19.2) | -27 (18.1)

43. Secondary Outcome: DBPC Period: Change From Baseline in Study 36-Item Short Form Health Survey Version 2 (SF-36v2) Physical Component Summary Score and Mental Component Summary Scores at Week 4, 8, 12, 16, 24, 32, 40 and 52
Description: The 36-Item Short-Form Health Survey (SF-36) was a standardized survey evaluating 8 aspects of functional health and well-being. These eight subscales were summarized as relating to either physical health or mental health. Physical component summary (PCS) was based primarily on physical functioning, role-physical, bodily pain, and general health scales and mental component summary (MCS) encompasses vitality, social functioning, role-emotional, and mental health scales. Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0 - 100 (100 = highest level of mental functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100 = highest level of physical functioning).
Time Frame: Baseline, Week 4, 8, 12, 16, 24, 32, 40 and 52
Population: Quality of Life analysis set included all randomized participants who had received at least 1 dose of IMP (Evobrutinib or placebo) and had at least 1 Baseline and 1 post baseline QoL assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 114 | 112 | 113
Units on a Scale
  Physical Component Summary Score at Week 4 | 1.2 (5.42) | 2.5 (7.40) | 3.5 (6.01) | 2.2 (5.86)
  Physical Component Summary Score at Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Physical Component Summary Score at Week 8 | 1.8 (6.35) | 3.5 (7.69) | 3.0 (6.61) | 2.2 (6.63)
  Physical Component Summary Score at Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Physical Component Summary Score at Week 12 | 2.4 (6.44) | 3.7 (7.71) | 4.2 (6.68) | 3.0 (6.99)
  Physical Component Summary Score at Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Physical Component Summary Score at Week 16 | 3.3 (7.04) | 4.0 (7.56) | 4.4 (5.81) | 3.4 (6.77)
  Physical Component Summary Score at Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Physical Component Summary Score at Week 24 | 3.4 (7.08) | 4.6 (7.57) | 5.4 (7.63) | 2.8 (7.15)
  Physical Component Summary Score at Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Physical Component Summary Score at Week 32 | 3.5 (8.03) | 3.8 (7.36) | 5.4 (7.24) | 3.8 (6.89)
  Physical Component Summary Score at Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Physical Component Summary Score at Week 40 | 4.2 (7.11) | 4.6 (7.97) | 5.7 (7.76) | 4.1 (8.59)
  Physical Component Summary Score at Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Physical Component Summary Score at Week 52 | 3.7 (8.32) | 5.4 (7.05) | 6.5 (8.58) | 4.8 (7.76)
  Mental Component Summary Score at Week 4 | 3.9 (9.38) | 1.7 (9.25) | 1.9 (7.93) | 2.4 (7.68)
  Mental Component Summary Score at Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Mental Component Summary Score at Week 8 | 2.5 (8.59) | 2.2 (8.81) | 1.6 (8.48) | 3.6 (9.04)
  Mental Component Summary Score at Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Mental Component Summary Score at Week 12 | 3.1 (10.07) | 3.1 (8.45) | 0.8 (10.39) | 2.9 (8.89)
  Mental Component Summary Score at Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Mental Component Summary Score at Week 16 | 3.6 (9.84) | 2.5 (8.39) | 2.8 (9.39) | 2.9 (9.13)
  Mental Component Summary Score at Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Mental Component Summary Score at Week 24 | 2.9 (9.75) | 2.4 (8.41) | 3.4 (9.68) | 2.7 (8.87)
  Mental Component Summary Score at Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Mental Component Summary Score at Week 32 | 3.5 (8.55) | 1.8 (9.51) | 2.8 (9.71) | 4.3 (9.03)
  Mental Component Summary Score at Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Mental Component Summary Score at Week 40 | 4.5 (8.81) | 1.5 (10.55) | 3.2 (9.81) | 4.0 (9.85)
  Mental Component Summary Score at Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Mental Component Summary Score at Week 52 | 3.8 (9.45) | 1.7 (9.91) | 3.9 (11.21) | 4.6 (9.80)

44. Secondary Outcome: DBPC Period: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire at Week 4, 8, 12, 16, 24, 32, 40 and 52
Description: The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L profile defines health in terms of mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has five levels: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, and 5: extreme problems. Responses were used to generate a weighted summary index (EQ-5D index), which ranges from 0 (dead) to 1.00 (perfect health). A higher score indicates better health and positive changes from baseline indicate improvement of health.
Time Frame: Baseline, Week 4, 8, 12, 16, 24, 32, 40, and 52
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 114 | 112 | 113
Units on a Scale
  Week 4 | 0.036 (0.1626) | 0.045 (0.1931) | 0.036 (0.1618) | 0.038 (0.1908)
  Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Week 8 | 0.034 (0.2164) | 0.064 (0.2505) | 0.046 (0.1842) | 0.061 (0.1603)
  Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Week 12 | 0.061 (0.2014) | 0.070 (0.2189) | 0.055 (0.1912) | 0.065 (0.1732)
  Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Week 16 | 0.083 (0.1818) | 0.072 (0.2252) | 0.067 (0.2287) | 0.056 (0.1738)
  Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Week 24 | 0.080 (0.1901) | 0.067 (0.2271) | 0.086 (0.2110) | 0.055 (0.1817)
  Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Week 32 | 0.083 (0.1758) | 0.067 (0.2262) | 0.075 (0.2009) | 0.071 (0.1941)
  Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Week 40 | 0.093 (0.1521) | 0.061 (0.1850) | 0.090 (0.1853) | 0.084 (0.2172)
  Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Week 52 | 0.096 (0.2092) | 0.078 (0.2197) | 0.102 (0.2224) | 0.096 (0.2051)

45. Secondary Outcome: DBPC Period: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Visual Analog Scale (VAS) at Week 4, 8, 12, 16, 24, 32, 40 and 52
Description: The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L profile defines health in terms of mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has five levels: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, and 5: extreme problems. The responses were used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 was the worst health you can imagine and 100 was the best health you can imagine.
Time Frame: Baseline, Week 4, 8, 12, 16, 24, 32, 40, and 52
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 114 | 112 | 113
Millimeter
  Week 4 | 3 (16.8) | 2 (19.0) | 4 (17.6) | 4 (18.2)
  Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Week 8 | 3 (18.8) | 6 (20.0) | 4 (14.5) | 6 (16.5)
  Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Week 12 | 5 (19.7) | 6 (17.4) | 5 (17.2) | 4 (16.8)
  Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Week 16 | 7 (19.3) | 5 (18.1) | 6 (18.5) | 4 (15.5)
  Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Week 24 | 7 (18.7) | 5 (18.4) | 9 (20.4) | 4 (17.3)
  Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Week 32 | 8 (17.2) | 4 (21.1) | 7 (17.8) | 7 (16.6)
  Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Week 40 | 8 (18.1) | 6 (18.1) | 10 (19.5) | 8 (18.9)
  Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Week 52 | 8 (19.9) | 8 (18.6) | 10 (21.3) | 10 (18.9)

46. Secondary Outcome: DBPC Period: Change From Baseline in Lupus Quality of Life (LupusQoL) Questionnaire Score at Week 4, 8, 12, 16, 24, 32, 40 and 52
Description: The Lupus QoL assessment is a 34 item questionnaire across 8 domains that is designed to find out how systemic lupus erythematosus (SLE) affects a participant's life. Domains include physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue. Participants indicate their responses on a 5-point Likert response format, where 4=never, 3=occasionally, 2= a good bit of the time, 1=most of the time, and 0=worst of the time. Summary scores can be calculated for all 8 domains. A LupusQoL score for each domain was reported on a 0 to 100 scale, with greater values indicating better health related QoL.
Time Frame: Baseline, Week 4, 8, 12, 16, 24, 32, 40, and 52
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 114 | 112 | 113
Units on a scale
  Physical Health Week 4 | 1.9 (12.58) | 4.7 (17.68) | 4.0 (14.04) | 3.5 (13.43)
  Physical Health Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Physical Health Week 8 | 2.8 (15.20) | 6.3 (19.94) | 3.8 (17.64) | 4.6 (14.69)
  Physical Health Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Physical Health Week 12 | 4.8 (16.75) | 6.7 (19.78) | 5.6 (15.95) | 5.7 (14.94)
  Physical Health Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Physical Health Week 16 | 6.6 (17.45) | 6.1 (18.71) | 7.4 (17.61) | 6.2 (15.59)
  Physical Health Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Physical Health Week 24 | 6.9 (17.17) | 7.2 (18.59) | 8.4 (20.47) | 6.1 (13.63)
  Physical Health Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Physical Health Week 32 | 5.7 (16.82) | 6.7 (19.45) | 9.4 (17.21) | 7.0 (16.21)
  Physical Health Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Physical Health Week 40 | 7.6 (15.32) | 8.2 (17.38) | 9.6 (19.10) | 7.1 (17.98)
  Physical Health Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Physical Health Week 52 | 7.1 (20.39) | 9.0 (18.44) | 11.6 (19.88) | 7.9 (18.73)
  Pain Week 4 | 3.6 (16.30) | 6.7 (21.81) | 9.0 (20.90) | 5.7 (16.26)
  Pain Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Pain Week 8 | 4.8 (18.71) | 9.9 (24.65) | 7.3 (21.76) | 6.7 (18.31)
  Pain Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Pain Week 12 | 7.5 (19.04) | 8.8 (24.00) | 9.8 (23.35) | 5.5 (14.73)
  Pain Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Pain Week 16 | 9.4 (18.58) | 8.3 (25.60) | 10.5 (26.33) | 6.9 (15.47)
  Pain Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Pain Week 24 | 9.4 (19.95) | 9.3 (24.31) | 13.0 (28.18) | 6.2 (17.02)
  Pain Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Pain Week 32 | 6.7 (23.74) | 9.2 (24.60) | 12.8 (22.87) | 8.7 (17.18)
  Pain Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Pain Week 40 | 11.0 (19.43) | 10.9 (23.68) | 15.3 (23.81) | 9.6 (20.51)
  Pain Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Pain Week 52 | 10.2 (21.37) | 12.9 (22.64) | 14.9 (26.11) | 9.6 (19.99)
  Planning Week 4 | 4.8 (20.14) | 4.9 (19.64) | 5.4 (24.30) | 4.6 (18.73)
  Planning Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Planning Week 8 | 5.5 (23.32) | 8.4 (23.25) | 5.8 (25.14) | 3.9 (22.98)
  Planning Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Planning Week 12 | 7.8 (23.58) | 5.8 (23.39) | 6.8 (25.74) | 5.1 (20.55)
  Planning Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Planning Week 16 | 8.3 (21.65) | 5.3 (24.12) | 6.5 (28.00) | 6.3 (22.91)
  Planning Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Planning Week 24 | 7.9 (22.92) | 8.1 (23.55) | 11.5 (29.08) | 5.6 (21.79)
  Planning Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Planning Week 32 | 6.5 (24.82) | 7.6 (22.66) | 9.9 (25.90) | 6.9 (22.07)
  Planning Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Planning Week 40 | 9.0 (20.69) | 7.8 (23.19) | 11.6 (26.17) | 8.0 (23.52)
  Planning Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Planning Week 52 | 9.9 (22.38) | 7.0 (23.12) | 9.9 (28.29) | 10.5 (21.59)
  Intimate Relationship Week 4: number analyzed (Participants) | 74 | 88 | 80 | 71
  Intimate Relationship Week 4 | 3.4 (26.11) | 1.6 (28.29) | 4.7 (24.06) | 3.2 (24.06)
  Intimate Relationship Week 8: number analyzed (Participants) | 70 | 81 | 75 | 61
  Intimate Relationship Week 8 | 8.2 (30.31) | 4.2 (28.44) | 9.7 (29.10) | 3.7 (18.73)
  Intimate Relationship Week 12: number analyzed (Participants) | 70 | 75 | 65 | 59
  Intimate Relationship Week 12 | 5.5 (27.31) | 4.7 (25.65) | 2.3 (30.37) | 6.4 (21.32)
  Intimate Relationship Week 16: number analyzed (Participants) | 60 | 72 | 69 | 53
  Intimate Relationship Week 16 | 8.8 (26.77) | 1.6 (30.76) | 3.8 (32.46) | 4.2 (22.99)
  Intimate Relationship Week 24: number analyzed (Participants) | 59 | 70 | 62 | 47
  Intimate Relationship Week 24 | 6.4 (30.12) | 2.1 (28.79) | 6.7 (30.76) | 5.3 (26.29)
  Intimate Relationship Week 32: number analyzed (Participants) | 54 | 66 | 54 | 52
  Intimate Relationship Week 32 | 2.5 (28.77) | 1.3 (31.78) | 6.5 (29.41) | 1.4 (27.86)
  Intimate Relationship Week 40: number analyzed (Participants) | 49 | 61 | 55 | 48
  Intimate Relationship Week 40 | 12.0 (27.59) | 6.6 (27.91) | 6.4 (32.53) | 7.8 (22.72)
  Intimate Relationship Week 52: number analyzed (Participants) | 51 | 60 | 49 | 45
  Intimate Relationship Week 52 | 7.4 (26.48) | 4.4 (28.36) | 8.4 (29.58) | 8.9 (24.52)
  Burden to Others Week 4 | 5.8 (23.83) | 5.2 (22.84) | 6.8 (24.85) | 2.2 (24.24)
  Burden to Others Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Burden to Others Week 8 | 5.6 (22.42) | 9.3 (27.17) | 5.7 (25.80) | 8.0 (25.79)
  Burden to Others Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Burden to Others Week 12 | 8.6 (25.86) | 6.7 (28.00) | 7.4 (25.93) | 7.3 (24.74)
  Burden to Others Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Burden to Others Week 16 | 11.8 (26.17) | 8.1 (23.32) | 6.7 (25.80) | 7.4 (24.30)
  Burden to Others Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Burden to Others Week 24 | 10.3 (28.68) | 9.0 (24.12) | 11.8 (27.15) | 5.8 (26.21)
  Burden to Others Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Burden to Others Week 32 | 10.6 (29.42) | 6.8 (24.09) | 9.6 (27.14) | 8.4 (28.21)
  Burden to Others Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Burden to Others Week 40 | 16.1 (25.07) | 12.4 (21.91) | 12.4 (28.74) | 12.1 (25.78)
  Burden to Others Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Burden to Others Week 52 | 15.3 (26.96) | 10.7 (22.13) | 13.0 (30.04) | 10.5 (25.89)
  Emotional Health Week 4 | 6.4 (15.37) | 4.7 (18.48) | 4.2 (18.45) | 1.8 (16.73)
  Emotional Health Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Emotional Health Week 8 | 4.5 (15.15) | 7.0 (19.26) | 2.3 (19.51) | 5.3 (15.53)
  Emotional Health Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Emotional Health Week 12 | 6.3 (17.23) | 7.6 (21.08) | 4.9 (20.99) | 4.7 (16.39)
  Emotional Health Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Emotional Health Week 16 | 8.3 (15.86) | 7.5 (19.59) | 7.4 (18.56) | 6.2 (18.32)
  Emotional Health Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Emotional Health Week 24 | 7.1 (17.31) | 5.6 (24.02) | 8.9 (20.97) | 4.3 (20.04)
  Emotional Health Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Emotional Health Week 32 | 6.3 (17.07) | 4.3 (23.55) | 9.0 (22.66) | 6.0 (20.56)
  Emotional Health Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Emotional Health Week 40 | 8.4 (16.08) | 8.3 (19.94) | 7.6 (21.52) | 6.7 (19.14)
  Emotional Health Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Emotional Health Week 52 | 8.5 (17.43) | 6.4 (21.31) | 8.2 (22.77) | 7.6 (18.80)
  Body Image Week 4: number analyzed (Participants) | 96 | 97 | 92 | 93
  Body Image Week 4 | 3.1 (17.70) | 8.4 (24.41) | 2.5 (24.60) | 4.0 (18.79)
  Body Image Week 8: number analyzed (Participants) | 90 | 92 | 91 | 85
  Body Image Week 8 | 5.7 (18.37) | 7.5 (23.40) | -1.3 (27.06) | 6.5 (17.30)
  Body Image Week 12: number analyzed (Participants) | 88 | 84 | 83 | 85
  Body Image Week 12 | 6.5 (18.57) | 7.1 (21.07) | 2.3 (26.86) | 6.6 (16.53)
  Body Image Week 16: number analyzed (Participants) | 84 | 82 | 85 | 81
  Body Image Week 16 | 6.7 (18.10) | 7.6 (23.11) | -0.4 (25.31) | 5.7 (20.39)
  Body Image Week 24: number analyzed (Participants) | 75 | 79 | 75 | 77
  Body Image Week 24 | 6.7 (20.84) | 10.2 (20.47) | 5.8 (27.31) | 6.7 (21.80)
  Body Image Week 32: number analyzed (Participants) | 71 | 76 | 68 | 73
  Body Image Week 32 | 5.1 (20.08) | 8.1 (23.71) | 3.3 (24.99) | 5.8 (21.54)
  Body Image Week 40: number analyzed (Participants) | 71 | 76 | 66 | 72
  Body Image Week 40 | 7.7 (14.11) | 8.2 (23.99) | 4.6 (26.67) | 9.0 (18.31)
  Body Image Week 52: number analyzed (Participants) | 74 | 68 | 66 | 67
  Body Image Week 52 | 6.6 (16.92) | 9.8 (21.46) | 5.1 (27.30) | 7.8 (21.56)
  Fatigue Week 4 | 4.4 (16.71) | 4.3 (18.98) | 6.2 (19.91) | 3.9 (17.08)
  Fatigue Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Fatigue Week 8 | 5.0 (19.22) | 7.1 (21.31) | 4.9 (20.61) | 4.5 (16.78)
  Fatigue Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Fatigue Week 12 | 6.7 (18.22) | 5.8 (21.30) | 7.3 (23.11) | 5.0 (16.08)
  Fatigue Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Fatigue Week 16 | 7.7 (17.61) | 6.6 (21.39) | 7.1 (24.16) | 4.1 (15.81)
  Fatigue Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Fatigue Week 24 | 7.5 (19.06) | 4.8 (23.34) | 9.0 (26.00) | 3.6 (14.20)
  Fatigue Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Fatigue Week 32 | 7.0 (19.20) | 3.7 (22.71) | 8.5 (22.96) | 4.1 (17.24)
  Fatigue Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Fatigue Week 40 | 11.3 (20.03) | 6.1 (25.28) | 11.0 (25.18) | 5.3 (16.73)
  Fatigue Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Fatigue Week 52 | 8.9 (21.15) | 4.5 (24.78) | 11.2 (22.56) | 6.7 (17.89)

47. Secondary Outcome: DBPC Period: Number of Participants With Patient Global Impression of Change (PGIC) Scale Score of Any Improvement, no Change and Any Worsening
Description: The PGIC is a self-rated scale that asks the participant to describe the change in activity limitations, symptoms, emotions, and overall quality of life (QoL) related to the participants painful condition on the following scale: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) and 7 (very much worse). Number of participants in the PGIC categories of any improvement (that is PGIC scale score 1, 2 or 3), no change (that is PGIC scale score 4) and any worsening (that is PGIC scale score 5, 6 or 7) are reported.
Time Frame: Week 4, 8, 12, 16, 24, 32, 40, and 52
Population: Quality of Life analysis set included all randomized participants who had received at least 1 dose of IMP (Evobrutinib or placebo) and had at least 1 Baseline and 1 post baseline QoL assessment. Here,"Number Analyzed" signified those participants who were evaluable at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 112 | 114 | 113 | 113
Participants
  Week 4: Any Improvement | 69 | 78 | 81 | 71
  Week 4: No Change | 33 | 27 | 23 | 34
  Week 4: Any Worsening | 8 | 9 | 8 | 8
  Week 4: Missing | 2 | 0 | 1 | 0
  Week 8: number analyzed (Participants) | 110 | 110 | 110 | 109
  Week 8: Any Improvement | 80 | 81 | 85 | 75
  Week 8: No Change | 22 | 18 | 19 | 28
  Week 8: Any Worsening | 5 | 9 | 5 | 3
  Week 8: Missing | 3 | 2 | 1 | 3
  Week 12: number analyzed (Participants) | 108 | 105 | 107 | 104
  Week 12: Any Improvement | 78 | 82 | 81 | 77
  Week 12: No Change | 23 | 13 | 15 | 20
  Week 12: Any Worsening | 5 | 7 | 7 | 4
  Week 12: Missing | 2 | 3 | 4 | 3
  Week 16: number analyzed (Participants) | 104 | 101 | 105 | 98
  Week 16: Any Improvement | 75 | 81 | 87 | 79
  Week 16: No Change | 23 | 13 | 16 | 15
  Week 16: Any Worsening | 3 | 7 | 2 | 2
  Week 16: Missing | 3 | 0 | 0 | 2
  Week 24: number analyzed (Participants) | 98 | 95 | 101 | 95
  Week 24: Any Improvement | 67 | 77 | 87 | 73
  Week 24: No Change | 23 | 12 | 7 | 17
  Week 24: Any Worsening | 6 | 6 | 5 | 5
  Week 24: Missing | 2 | 0 | 2 | 0
  Week 32: number analyzed (Participants) | 91 | 91 | 95 | 89
  Week 32: Any Improvement | 70 | 70 | 80 | 72
  Week 32: No Change | 16 | 15 | 8 | 13
  Week 32: Any Worsening | 4 | 6 | 5 | 3
  Week 32: Missing | 1 | 0 | 2 | 1
  Week 40: number analyzed (Participants) | 89 | 89 | 93 | 87
  Week 40: Any Improvement | 67 | 69 | 80 | 73
  Week 40: No Change | 19 | 12 | 7 | 9
  Week 40: Any Worsening | 2 | 8 | 4 | 4
  Week 40: Missing | 1 | 0 | 2 | 1
  Week 52: number analyzed (Participants) | 88 | 89 | 90 | 85
  Week 52: Any Improvement | 66 | 64 | 76 | 64
  Week 52: No Change | 14 | 18 | 6 | 13
  Week 52: Any Worsening | 6 | 1 | 5 | 4
  Week 52: Missing | 2 | 6 | 3 | 4

48. Secondary Outcome: DBPC Period: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 4, 8, 12, 16, 24, 32, 40 and 52
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assess self reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse possible score) to 52 (best score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 4, 8, 12, 16, 24, 32, 40, and 52
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 110 | 114 | 112 | 113
Units on a scale
  Week 4 | 3 (8.0) | 2 (7.8) | 4 (9.1) | 3 (7.7)
  Week 8: number analyzed (Participants) | 107 | 108 | 109 | 106
  Week 8 | 3 (8.7) | 3 (8.3) | 3 (9.1) | 5 (8.2)
  Week 12: number analyzed (Participants) | 106 | 102 | 103 | 101
  Week 12 | 3 (10.0) | 4 (9.7) | 3 (9.7) | 4 (8.1)
  Week 16: number analyzed (Participants) | 101 | 101 | 105 | 96
  Week 16 | 4 (9.8) | 3 (9.8) | 4 (10.2) | 3 (8.4)
  Week 24: number analyzed (Participants) | 96 | 95 | 99 | 95
  Week 24 | 3 (9.9) | 4 (8.5) | 5 (10.3) | 3 (7.5)
  Week 32: number analyzed (Participants) | 90 | 91 | 93 | 88
  Week 32 | 4 (9.6) | 4 (9.5) | 5 (9.7) | 4 (6.8)
  Week 40: number analyzed (Participants) | 88 | 89 | 91 | 86
  Week 40 | 4 (8.8) | 3 (8.6) | 6 (9.9) | 4 (8.5)
  Week 52: number analyzed (Participants) | 86 | 84 | 87 | 82
  Week 52 | 4 (9.9) | 4 (7.9) | 5 (9.7) | 5 (8.7)

49. Secondary Outcome: DBPC Period: Number of Participants With Change From Baseline in Prednisone Equivalent Corticosteroid (CS) Dose by >=25% to a Dose of <=7.5 Milligram Per Day (mg/Day), With no BILAG A or 2B Flare in Disease Activity at Week 52
Description: BILAG A or 2B flare is defined as at least one BILAG A grade or two BILAG B grade in any organ system due to items that are new or worse, compared to the BILAG evaluation at the previous visit, during the 52 week treatment period. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to systemic lupus erythematosus (SLE), divided into 9 organ systems. For each organ system based on alphabetic score: A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected.
Time Frame: Baseline and Week 52
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 68 | 68 | 70 | 71
Participants | 19 | 23 | 20 | 21
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; Rate difference = 5.9, 95% CI 2-sided [-9.7 to 21.2]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; Rate Difference = 0.6, 95% CI 2-sided [-14.5 to 15.6]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; Rate difference = 1.6, 95% CI 2-sided [-13.5 to 16.6]

50. Secondary Outcome: DBPC Period: Change From Baseline to Week 52 in Prednisone Equivalent Corticosteroid (CS) Daily Dose at at Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: Change From Baseline in Prednisone-equivalent CS Daily Dose at Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 were reported.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. . Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Milligram (mg)
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 113 | 113 | 116 | 114
Milligram (mg)
  Week 1: number analyzed (Participants) | 48 | 58 | 60 | 52
  Week 1 | 0.21 (1.443) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Week 2 | 0.10 (1.206) | -0.07 (0.524) | 0.00 (0.000) | -0.13 (1.405)
  Week 4: number analyzed (Participants) | 111 | 113 | 115 | 111
  Week 4 | 0.01 (1.267) | -0.45 (2.879) | -0.04 (0.739) | -0.15 (1.428)
  Week 6: number analyzed (Participants) | 57 | 47 | 55 | 55
  Week 6 | -1.07 (3.563) | -0.64 (3.275) | -0.59 (2.095) | -0.70 (3.484)
  Week 8: number analyzed (Participants) | 108 | 110 | 110 | 105
  Week 8 | -0.57 (2.588) | -1.24 (3.915) | -1.09 (3.640) | -1.02 (3.422)
  Week 10: number analyzed (Participants) | 55 | 49 | 61 | 55
  Week 10 | -1.43 (3.985) | -2.04 (5.146) | -1.56 (4.137) | -2.50 (4.971)
  Week 12: number analyzed (Participants) | 107 | 102 | 107 | 99
  Week 12 | -1.26 (3.260) | -1.85 (4.158) | -1.73 (4.574) | -1.97 (4.150)
  Week 14: number analyzed (Participants) | 60 | 51 | 63 | 57
  Week 14 | -2.00 (4.569) | -2.70 (5.428) | -1.87 (4.489) | -2.76 (5.125)
  Week 16: number analyzed (Participants) | 102 | 101 | 104 | 97
  Week 16 | -1.67 (4.427) | -2.70 (4.955) | -2.47 (5.365) | -2.40 (4.535)
  Week 20: number analyzed (Participants) | 98 | 94 | 101 | 94
  Week 20 | -1.94 (4.054) | -2.82 (4.905) | -2.64 (5.489) | -2.53 (4.727)
  Week 24: number analyzed (Participants) | 93 | 95 | 99 | 91
  Week 24 | -1.99 (4.228) | -2.64 (5.066) | -2.61 (5.568) | -2.34 (5.330)
  Week 28: number analyzed (Participants) | 92 | 91 | 97 | 89
  Week 28 | -2.23 (4.439) | -2.97 (4.981) | -3.07 (6.068) | -2.46 (5.371)
  Week 32: number analyzed (Participants) | 92 | 90 | 95 | 88
  Week 32 | -2.45 (4.584) | -3.13 (5.193) | -3.18 (6.161) | -2.44 (5.347)
  Week 36: number analyzed (Participants) | 90 | 90 | 95 | 87
  Week 36 | -2.42 (4.835) | -3.31 (5.327) | -3.18 (6.136) | -2.37 (5.445)
  Week 40: number analyzed (Participants) | 90 | 90 | 92 | 86
  Week 40 | -2.08 (6.149) | -3.21 (5.280) | -3.24 (6.218) | -2.67 (5.202)
  Week 44: number analyzed (Participants) | 89 | 90 | 92 | 85
  Week 44 | -2.42 (4.833) | -3.21 (5.280) | -3.27 (6.254) | -2.56 (5.121)
  Week 48: number analyzed (Participants) | 86 | 89 | 91 | 84
  Week 48 | -2.38 (4.895) | -3.22 (5.310) | -3.37 (6.265) | -2.62 (5.136)
  Week 52: number analyzed (Participants) | 99 | 100 | 100 | 96
  Week 52 | -1.70 (5.470) | -2.94 (5.534) | -3.09 (5.981) | -2.63 (5.673)

51. Secondary Outcome: DBPC Period: Number of Participants With Reduction From Baseline in Prednisone Equivalent Corticosteroid (CS) Daily Dose by > 0 to 25%, >25% to 50%, >50% to 100% or an Increase at Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Description: Number of Participants With Reduction From Baseline in Prednisone-equivalent Corticosteroid (CS) Daily Dose by > 0 to 25%, >25% to 50%, >50% to 100% or an Increase at Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 were reported.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants
  Reduction of dose by >0-25% Week 1 | 0 | 0 | 0 | 0
  Reduction of dose by >0-25% Week 2 | 1 | 2 | 0 | 0
  Reduction of dose by >0-25% Week 4 | 1 | 5 | 2 | 1
  Reduction of dose by >0-25% Week 6 | 3 | 4 | 3 | 4
  Reduction of dose by >0-25% Week 8 | 6 | 6 | 5 | 6
  Reduction of dose by >0-25% Week 10 | 0 | 3 | 4 | 5
  Reduction of dose by >0-25% Week 12 | 5 | 11 | 8 | 6
  Reduction of dose by >0-25% Week 14 | 2 | 2 | 4 | 5
  Reduction of dose by >0-25% Week 16 | 5 | 10 | 5 | 6
  Reduction of dose by >0-25% Week 20 | 5 | 10 | 5 | 5
  Reduction of dose by >0-25% Week 24 | 4 | 10 | 5 | 5
  Reduction of dose by >0-25% Week 28 | 2 | 8 | 5 | 4
  Reduction of dose by >0-25% Week 32 | 1 | 7 | 4 | 3
  Reduction of dose by >0-25% Week 36 | 1 | 5 | 4 | 3
  Reduction of dose by >0-25% Week 40 | 1 | 5 | 3 | 3
  Reduction of dose by >0-25% Week 44 | 1 | 5 | 3 | 3
  Reduction of dose by >0-25% Week 48 | 0 | 5 | 4 | 3
  Reduction of dose by >0-25% Week 52 | 1 | 5 | 4 | 4
  Reduction of dose by >25- 50% Week 1 | 0 | 0 | 0 | 0
  Reduction of dose by >25- 50% Week 2 | 0 | 0 | 0 | 0
  Reduction of dose by >25- 50% Week 4 | 1 | 2 | 1 | 0
  Reduction of dose by >25- 50% Week 6 | 4 | 1 | 2 | 0
  Reduction of dose by >25- 50% Week 8 | 5 | 9 | 6 | 5
  Reduction of dose by >25- 50% Week 10 | 7 | 6 | 4 | 10
  Reduction of dose by >25- 50% Week 12 | 14 | 9 | 10 | 15
  Reduction of dose by >25- 50% Week 14 | 7 | 6 | 2 | 8
  Reduction of dose by >25- 50% Week 16 | 16 | 12 | 9 | 16
  Reduction of dose by >25- 50% Week 20 | 13 | 11 | 8 | 14
  Reduction of dose by >25- 50% Week 24 | 12 | 9 | 8 | 13
  Reduction of dose by >25- 50% Week 28 | 14 | 12 | 9 | 16
  Reduction of dose by >25- 50% Week 32 | 15 | 11 | 8 | 16
  Reduction of dose by >25- 50% Week 36 | 15 | 13 | 6 | 15
  Reduction of dose by >25- 50% Week 40 | 15 | 15 | 6 | 16
  Reduction of dose by >25- 50% Week 44 | 15 | 15 | 6 | 16
  Reduction of dose by >25- 50% Week 48 | 15 | 14 | 6 | 17
  Reduction of dose by >25- 50% Week 52 | 16 | 12 | 7 | 17
  Reduction of dose by >50-100% Week 1 | 0 | 0 | 0 | 0
  Reduction of dose by >50-100% Week 2 | 0 | 0 | 0 | 1
  Reduction of dose by >50-100% Week 4 | 0 | 1 | 0 | 1
  Reduction of dose by >50-100% Week 6 | 1 | 1 | 0 | 1
  Reduction of dose by >50-100% Week 8 | 1 | 3 | 4 | 3
  Reduction of dose by >50-100% Week 10 | 2 | 3 | 3 | 4
  Reduction of dose by >50-100% Week 12 | 1 | 6 | 6 | 6
  Reduction of dose by >50-100% Week 14 | 5 | 6 | 7 | 7
  Reduction of dose by >50-100% Week 16 | 5 | 13 | 13 | 9
  Reduction of dose by >50-100% Week 20 | 7 | 13 | 14 | 11
  Reduction of dose by >50-100% Week 24 | 7 | 14 | 13 | 11
  Reduction of dose by >50-100% Week 28 | 9 | 14 | 15 | 11
  Reduction of dose by >50-100% Week 32 | 11 | 16 | 16 | 12
  Reduction of dose by >50-100% Week 36 | 10 | 17 | 18 | 11
  Reduction of dose by >50-100% Week 40 | 10 | 15 | 18 | 11
  Reduction of dose by >50-100% Week 44 | 10 | 15 | 18 | 10
  Reduction of dose by >50-100% Week 48 | 9 | 15 | 19 | 10
  Reduction of dose by >50-100% Week 52 | 9 | 17 | 19 | 12
  Increased from Baseline Week 1 | 1 | 0 | 0 | 0
  Increased from Baseline Week 2 | 2 | 0 | 0 | 0
  Increased from Baseline Week 4 | 2 | 1 | 1 | 0
  Increased from Baseline Week 6 | 1 | 1 | 0 | 0
  Increased from Baseline Week 8 | 2 | 1 | 1 | 0
  Increased from Baseline Week 10 | 1 | 1 | 0 | 0
  Increased from Baseline Week 12 | 1 | 1 | 1 | 0
  Increased from Baseline Week 14 | 1 | 0 | 0 | 0
  Increased from Baseline Week 16 | 1 | 1 | 1 | 0
  Increased from Baseline Week 20 | 0 | 0 | 0 | 0
  Increased from Baseline Week 24 | 0 | 0 | 0 | 0
  Increased from Baseline Week 28 | 0 | 0 | 0 | 1
  Increased from Baseline Week 32 | 0 | 0 | 0 | 1
  Increased from Baseline Week 36 | 0 | 0 | 0 | 1
  Increased from Baseline Week 40 | 1 | 0 | 0 | 1
  Increased from Baseline Week 44 | 0 | 0 | 0 | 1
  Increased from Baseline Week 48 | 0 | 0 | 0 | 1
  Increased from Baseline Week 52 | 2 | 0 | 0 | 2

52. Secondary Outcome: DBPC Period: Cumulative Prednisone Equivalent Corticosteroid (CS) Dose at Week 52
Description: Cumulative Prednisone-equivalent Corticosteroid (CS) Dose was calculated at Week 52.
Time Frame: Week 52
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Milligrams | 2267.66 (1507.652) | 2209.46 (1922.557) | 2137.70 (1618.688) | 2205.56 (1737.092)

53. Secondary Outcome: DBPC Period: Number of Participants With a Sustained Reduction of Oral Corticosteroids (OCS) Dose to 7.5 mg Prednisone Equivalent Per Day or Less With Response Based on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Week 52
Description: as for outcome 31
Time Frame: Week 52
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 56 | 59 | 63 | 57
Participants | 43 | 45 | 43 | 41
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.7728, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.46 to 2.82]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.3314, Regression, Logistic; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.28 to 1.54]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.7205, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.36 to 2.04]

54. Secondary Outcome: DBPC Period: Number of Participants With a Sustained Reduction of Oral Corticosteroids (OCS) Dose to 7.5 mg Prednisone Equivalent Per Day or Less With Response Based on Systemic Lupus Erythematosus Responder Index 6 (SRI-6) at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "overall number of participants analyzed" signifies those participants who achieved SLEDAI-2K total score >= 10 at screening (HDA participants) and evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 27 | 28 | 35 | 24
Participants | 18 | 19 | 23 | 15
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.8364, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.35 to 3.71]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.8287, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.37 to 3.45]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.7621, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.35 to 4.16]

55. Secondary Outcome: DBPC Period: Number of Participants With a Sustained Reduction of Oral Corticosteroids (OCS) Dose to 7.5 mg Prednisone Equivalent Per Day or Less With Response Based on SRI-4 at Week 52 in Serologically Active Subgroup
Description: SRI-4 response was defined as greater than or equal to (>=) 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score, no worsening (less than 10 percent increase) from baseline in Physician's Global Assessment of Disease Activity (PGA) and no treatment failure. SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms, or laboratory parameters related to Systemic Lupus Erythematosus (SLE), divided into 9 organ systems. For each organ system A=severe disease, B=moderate disease, C=mild stable disease, D=inactive, but previously active, E=inactive and never affected. The PGA assess disease activity on a visual analogue scale = from very well(0)-very poor(100).
Time Frame: Week 52
Population: The mITT analysis set included all randomized participants who had received at least one dose of IMP (Evobrutinib or placebo) and have at least one Baseline and one post Baseline disease assessment among the following: SFI, SLEDAI 2K, PGA, BILAG 2004, CLASI. Here, "Overall Number of Participants Analyzed" signifies those participants with positive antidsDNA and/or low complement levels at screening (Serologically active subgroup) and evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 26 | 33 | 32 | 34
Participants | 21 | 25 | 22 | 25
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.8464, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.23 to 3.31]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.4170, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.16 to 2.12]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.9988, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.27 to 3.74]

56. Secondary Outcome: DBPC Period: Number of Participants With Lupus Low Disease Activity State (LLDAS) at Week 52
Description: Lupus low disease activity state will be measured as: SLEDAI-2K <= 4; No activity in any major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever); No new features of disease activity compared with the previous assessment; Prednisone-equivalent <= 7.5 milligram per day; Unchanged background immunosuppressive therapy.
Time Frame: Week 52
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID
Number analyzed (Participants) | 114 | 115 | 116 | 114
Participants | 29 | 32 | 35 | 29
Statistical Analysis 1: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 25 mg QD; Test type: Superiority; p = 0.6970, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.62 to 2.04]
Statistical Analysis 2: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 75 mg QD; Test type: Superiority; p = 0.3234, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.75 to 2.42]
Statistical Analysis 3: Comparison: DBPC Period: Placebo vs DBPC Period: M2951 50 mg BID; Test type: Superiority; p = 0.9846, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.54 to 1.82]

ADVERSE EVENTS:
Time Frame: Double-Blind Placebo-Controlled: Baseline up to Week 56 Long-Term Extension: Up to Week 108
Arm/Group | DBPC Period: Placebo | DBPC Period: M2951 25 mg QD | DBPC Period: M2951 75 mg QD | DBPC Period: M2951 50 mg BID | LTE: Placebo/ M2951 50 mg BID | LTE Period: M2951 25 mg QD/ M2951 50 mg BID | LTE Period: M2951 75 mg QD/ M2951 50 mg BID | LTE: M2951 50 mg BID/ M2951 50 mg BID
All-Cause Mortality (participants affected / at risk) | 0/117 | 1/118 | 1/117 | 0/117 | 0/62 | 0/69 | 0/80 | 0/72
Serious Adverse Events (participants affected / at risk) | 10/117 | 13/118 | 11/117 | 9/117 | 5/62 | 5/69 | 5/80 | 7/72
Other Adverse Events (participants affected / at risk) | 76/117 | 85/118 | 75/117 | 78/117 | 22/62 | 34/69 | 35/80 | 23/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBPC Period: Placebo (N=117) | DBPC Period: M2951 25 mg QD (N=118) | DBPC Period: M2951 75 mg QD (N=117) | DBPC Period: M2951 50 mg BID (N=117) | LTE: Placebo/ M2951 50 mg BID (N=62) | LTE Period: M2951 25 mg QD/ M2951 50 mg BID (N=69) | LTE Period: M2951 75 mg QD/ M2951 50 mg BID (N=80) | LTE: M2951 50 mg BID/ M2951 50 mg BID (N=72)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis lupus (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lupus enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Campylobacter sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subperiosteal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBPC Period: Placebo (N=117) | DBPC Period: M2951 25 mg QD (N=118) | DBPC Period: M2951 75 mg QD (N=117) | DBPC Period: M2951 50 mg BID (N=117) | LTE: Placebo/ M2951 50 mg BID (N=62) | LTE Period: M2951 25 mg QD/ M2951 50 mg BID (N=69) | LTE Period: M2951 75 mg QD/ M2951 50 mg BID (N=80) | LTE: M2951 50 mg BID/ M2951 50 mg BID (N=72)
Lymphopenia (Blood and lymphatic system disorders) | 9 | 4 | 6 | 2 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 6 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 12 | 17 | 10 | 3 | 5 | 7 | 2
Nausea (Gastrointestinal disorders) | 7 | 8 | 9 | 5 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 9 | 8 | 3 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6 | 8 | 5 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 3 | 5 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 6 | 3 | 4 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 5 | 7 | 9 | 7 | 4 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 16 | 21 | 26 | 21 | 4 | 7 | 7 | 6
Nasopharyngitis (Infections and infestations) | 8 | 13 | 15 | 7 | 5 | 5 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 12 | 15 | 6 | 8 | 3 | 6 | 3 | 0
Pharyngitis (Infections and infestations) | 8 | 5 | 4 | 4 | 0 | 3 | 6 | 1
Gastroenteritis (Infections and infestations) | 6 | 4 | 2 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 6 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 8 | 6 | 6 | 5 | 4 | 1 | 2
Lipase increased (Investigations) | 2 | 4 | 6 | 6 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 8 | 3 | 4 | 3 | 4 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 6 | 4 | 4 | 7 | 3 | 3 | 1 | 4
Amylase increased (Investigations) | 5 | 2 | 4 | 8 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 3 | 3 | 3 | 6 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5 | 9 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 20 | 17 | 19 | 17 | 1 | 7 | 2 | 5
Dizziness (Nervous system disorders) | 3 | 5 | 4 | 6 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 6 | 4 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 3

LIMITATIONS AND CAVEATS:
Primary and Secondary endpoints were planned to be analyze only for Double-Blind Placebo-controlled period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02975336/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02975336/SAP_001.pdf